CLINICAL TRIAL: NCT06367621
Title: Retrospective Evaluation of Diagnostic Specificity and Sensitivity for iStatis Syphilis Ab Test at the Point-Of-Care Sites
Brief Title: Retrospective Study of iStatis Syphilis Ab Test (POC)
Status: Completed | Type: Observational
Sponsor: bioLytical Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: CLS-015C
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Syphilis; Syphilis Infection
Keywords: diagnostic kit; diagnostic devices; lateral flow device test; syphilis rapid test; syphilis point of care tests; iStatis Syphilis Antibody Test
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Retrospective samples are used for testing with the investigational device as well as reference testing. All remaining samples are retained per site policy and procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- iStatis Syphilis Antibody Test diagnostic device: Bio-banked plasma and serum samples available to Epicentre Health Research will be used for testing on iStatis Syphilis Antibody Test device.
  Interventions: Device: iStatis Syphilis Antibody Test
- Reference test: Either serum or plasma samples were tested with Abbott Architect Syphilis Tp (EDA) and MD Macro-Vue Particle Agglutination (RPR)/Serodia Particle Agglutination (TPPA) where applicable

INTERVENTIONS:
Device: iStatis Syphilis Antibody Test — 1500 stored samples (plasma/serum) will be tested in a routine testing environment using the iStatis Syphilis Antibody Test diagnostic device. Results of tests will not be used for patient management decisions (observaltional).
  Groups: iStatis Syphilis Antibody Test diagnostic device

SUMMARY:
The purpose of this retrospective clinical trial is to establish the clinical performance of the iStatis Syphilis AbTest. The data will be used to demonstrate the product is safe and effective for its intended use. The data obtained will be used in the application for CE certification under In Vitro Diagnostic Medical Device Regulation (IVDR) and World Health Organization (WHO) prequalification.

DETAILED DESCRIPTION:
The objectives of this study are to establish the diagnostic sensitivity and diagnostic specificity of the iStatis Syphilis Ab Test. Left-over samples stored at -80ᵒC from the previous trials conducted by Epicentre will be used for this study. The samples are tested in a routine testing environment. Serum samples were tested for evidence of syphilis infection using a non-treponemal Rapid Plasma Reagin (RPR) assay. All reactive samples were further tested quantitatively.

ELIGIBILITY:
Inclusion Criteria:

1. Anti-Tp negative samples:

   -Stored at ≤ -80°C.
2. Anti-Tp negative samples - pregnant women:

   * Samples from pregnant women, 1st and multipara
   * Samples found negative or false reactive for anti-Tp assay with the reference method.
   * Stored at ≤ -80°C.
3. Anti-Tp positive samples:

   * Samples screened with Abbott Architect Syphilis Tp and confirmed positive with BD Macro-Vue Particle Agglutination (RPR) and Serodia Particle Agglutination (TPPA).
   * Stored at ≤ -80°C.
4. Anti-Tp positive samples - pregnant women:

   * Samples from pregnant women
   * Samples screened with Abbott Architect Syphilis Tp and confirmed positive with BD Macro-Vue Particle Agglutination (RPR) and Serodia Particle Agglutination (TPPA).
   * Stored at ≤ -80°C.

Exclusion Criteria:

* N/A

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective cross-sectional study on left-over samples stored at -80°C from previous trials conducted by Epicentre Heath Research.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the iStatis Syphilis Ab Test | 8 weeks
  To estimate the diagnostic specificity and diagnostic sensitivity of the iStatis Syphilis Antibody Test in detecting anti-Tp in plasma and serum

CONTACTS AND LOCATIONS:
Locations (1):
- Epicentre Health Research, Hillcrest, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No